CLINICAL TRIAL: NCT02728635
Title: Epigenetic Regulation of Human Adipose Tissue Distribution
Acronym: Eiffel 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Sanford-Burnham Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMDFH 869496
Record Dates: First submitted 2016-03-24; First posted 2016-04-05 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Adipose tissue, epigenetic, abdominal gluteal fat
MeSH Terms: conditions — Obesity | interventions — Absorptiometry, Photon; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A- Women- Healthy 'pears' (Active Comparator): This group will consist of healthy women with a BMI between 23 and 35 kg/m2 as a waist-to-hip ratio of 0.78 or less.
  Interventions: Other: Dual-energy X-ray absorptiometry (DEXA)/ Magnetic resonance imaging (MRI) and Magnetic resonance spectroscopy (MRS); Procedure: Adipose tissue biopsies; Other: FSIGTT/ RMR
- Group B- Women- Healthy 'apples' (Active Comparator): The group will consist of healthy women with a BMI between 23 and 35 kg/m2 as a waist-to-hip ratio of 0.85 or more.
  Interventions: Other: Dual-energy X-ray absorptiometry (DEXA)/ Magnetic resonance imaging (MRI) and Magnetic resonance spectroscopy (MRS); Procedure: Adipose tissue biopsies; Other: FSIGTT/ RMR
- Group C- Men- Healthy 'apples' (Active Comparator): The group will consist of men with a BMI between 23 and 35 kg/m2.
  Interventions: Other: Dual-energy X-ray absorptiometry (DEXA)/ Magnetic resonance imaging (MRI) and Magnetic resonance spectroscopy (MRS); Procedure: Adipose tissue biopsies; Other: FSIGTT/ RMR

INTERVENTIONS:
Other: Dual-energy X-ray absorptiometry (DEXA)/ Magnetic resonance imaging (MRI) and Magnetic resonance spectroscopy (MRS) — A DEXA scan for body composition will also be completed. After a MRI safety screening a whole body MRI for the volumetric measurement of visceral fat, subcutaneous fat, liver, kidneys, heart, brain, skeletal muscle and intramuscular adipose tissue (IMAT) and hepatic lipid by MRS will be performed. Whole body imaging will include low resolution positioning images, followed by several sets of 3D images which will be digitally connected to create a 3D image the entire length of the body. The liver spectroscopy will be performed using PRESS (point resolved spectroscopy) and STEAM (Stimulated Echo Acquisition Mode) sequence during the same imaging session, using the whole body images for positioning.
Procedure: Adipose tissue biopsies — Two biopsies will be performed to collect fat tissue from the abdomen and thigh region.
Other: FSIGTT/ RMR — Insertion of two intravenous (IV) catheters for performing a Frequently Sampled Intravenous Glucose Tolerance Test (FSIGTT) to measure the acute insulin response to glucose (AIRg) and insulin sensitivity (Si) will be performed. Resting metabolic rate (RMR) will be used to measure metabolic flexibility. Point of care blood glucose measurements will be taken frequently to ensure safety.

SUMMARY:
The purpose of this study is to collect data to help researchers better understand the different ways that women or men store fat (apple shape versus pear shape).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years inclusive;
* BMI 23-35 kg/m2 inclusive;
* HbA1C <6.0%;
* Weight stable (± 3 kg) during the 3 months prior to enrollment;
* Women must be > 9 months post-partum;
* Able to provide written, informed consent.

Exclusion Criteria:

* Postmenopausal women
* Women with an oophorectomy
* Fasting plasma glucose > 126 mg/dL, or diagnosis with Type 2 Diabetes (T2DM)
* Untreated or symptomatic thyroid disease.
* Aminotransferase or aspartate aminotransferase > 3x upper limit of laboratory reference range, or known diagnosis of liver disease.
* Creatinine > 2x upper limit of laboratory reference range, or known diagnosis of kidney disease.
* Uncontrolled hypertension (BP > 140 systolic or > 90 diastolic)
* New onset (<3 months on a stable regime) use of oral contraceptives or hormone replacement therapy.
* History of drug or alcohol abuse (> 3 drinks per day) within the last 5 years, or psychiatric disease prohibiting adherence to study protocol. Current drug use may be determine by plasma or urine drug screens.
* History of cancer within the last 5 years (skin cancers, with the exception of melanoma, may be acceptable).
* History of organ transplant.
* Myocardial Infarction within the last 6 months.
* Current treatment with blood thinners or antiplatelet medications that cannot be safely stopped for biopsy and testing procedures.
* History of HIV, active Hepatitis B or C or tuberculosis
* Presence of clinically significant abnormalities on EKG.
* Current smokers (smoking within the past 3 months).
* Use of any medications known to influence glucose, fat and/or energy metabolism within the last 3 months (eg. growth hormone therapy, glucocorticoids [steroids], etc.)
* Other chronic or acute illness that might affect study results / interpretation in the opinion of the clinical
* Other items related to procedural risk (outlined below) such as bleeding disorder, claustrophobia, etc.
* Elevated high sensitivity c-reactive protein or known active infection.
* There are some implants which are MR compatible (safe) but would cause artifacts which could obscure our ability to measure an organ, e.g. full braces may negate the ability to measure brain size.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Epigenetic marks in abdominal vs gluteal subcutaneous adipose tissue and adipocytes | 6 weeks
  The preadipocytes obtained from biopsies of Abdominal Fat and Gluteofemoral Fat from patients in the 'pears' woman, 'apple' women and men will be cultured by our standard methods in proliferative medium followed by our standard protocol for differentiation into mature adipocytes. We propose to evaluate samples from 3 individuals from each Group to identify a large number of differentially regulated regions genome wide. All the data obtained in vitro in culture cells will be compared with the data obtained from RNA and chromatin isolated from the whole tissue Abdominal fat and Gluteofemoral fat biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] McAllister EJ, Dhurandhar NV, Keith SW, Aronne LJ, Barger J, Baskin M, Benca RM, Biggio J, Boggiano MM, Eisenmann JC, Elobeid M, Fontaine KR, Gluckman P, Hanlon EC, Katzmarzyk P, Pietrobelli A, Redden DT, Ruden DM, Wang C, Waterland RA, Wright SM, Allison DB. Ten putative contributors to the obesity epidemic. Crit Rev Food Sci Nutr. 2009 Nov;49(10):868-913. doi: 10.1080/10408390903372599. PMID 19960394
- [Background] Roberson L, Shaharyar S, Aneni E, Freitas W, Blaha M, Agatston A, Blumenthal R, Santos RD, Feiz H, Nasir K, Sposito A. The prevalence of the metabolically healthy obese phenotype in an aging population and its association with subclinical cardiovascular disease: The Brazilian study on healthy aging. Diabetol Metab Syndr. 2014 Nov 7;6(1):121. doi: 10.1186/1758-5996-6-121. eCollection 2014. PMID 25411583
- [Background] Roberson LL, Aneni EC, Maziak W, Agatston A, Feldman T, Rouseff M, Tran T, Blaha MJ, Santos RD, Sposito A, Al-Mallah MH, Blankstein R, Budoff MJ, Nasir K. Beyond BMI: The "Metabolically healthy obese" phenotype & its association with clinical/subclinical cardiovascular disease and all-cause mortality -- a systematic review. BMC Public Health. 2014 Jan 8;14:14. doi: 10.1186/1471-2458-14-14. PMID 24400816
- [Background] de Koning L, Merchant AT, Pogue J, Anand SS. Waist circumference and waist-to-hip ratio as predictors of cardiovascular events: meta-regression analysis of prospective studies. Eur Heart J. 2007 Apr;28(7):850-6. doi: 10.1093/eurheartj/ehm026. Epub 2007 Apr 2. PMID 17403720
- [Background] Qiao Q, Nyamdorj R. Is the association of type II diabetes with waist circumference or waist-to-hip ratio stronger than that with body mass index? Eur J Clin Nutr. 2010 Jan;64(1):30-4. doi: 10.1038/ejcn.2009.93. Epub 2009 Sep 2. PMID 19724291
- [Background] Yusuf S, Hawken S, Ounpuu S, Bautista L, Franzosi MG, Commerford P, Lang CC, Rumboldt Z, Onen CL, Lisheng L, Tanomsup S, Wangai P Jr, Razak F, Sharma AM, Anand SS; INTERHEART Study Investigators. Obesity and the risk of myocardial infarction in 27,000 participants from 52 countries: a case-control study. Lancet. 2005 Nov 5;366(9497):1640-9. doi: 10.1016/S0140-6736(05)67663-5. PMID 16271645
- [Background] VAGUE J. The degree of masculine differentiation of obesities: a factor determining predisposition to diabetes, atherosclerosis, gout, and uric calculous disease. Am J Clin Nutr. 1956 Jan-Feb;4(1):20-34. doi: 10.1093/ajcn/4.1.20. No abstract available. PMID 13282851
- [Background] Vague J. Sexual differentiation. A determinant factor of the forms of obesity. 1947. Obes Res. 1996 Mar;4(2):201-3. doi: 10.1002/j.1550-8528.1996.tb00535.x. No abstract available. PMID 8681056
- [Background] Santosa S, Jensen MD. Why are we shaped differently, and why does it matter? Am J Physiol Endocrinol Metab. 2008 Sep;295(3):E531-5. doi: 10.1152/ajpendo.90357.2008. Epub 2008 May 20. PMID 18492764
- [Background] Fu J, Hofker M, Wijmenga C. Apple or pear: size and shape matter. Cell Metab. 2015 Apr 7;21(4):507-8. doi: 10.1016/j.cmet.2015.03.016. PMID 25863240
- [Background] Manolopoulos KN, Karpe F, Frayn KN. Gluteofemoral body fat as a determinant of metabolic health. Int J Obes (Lond). 2010 Jun;34(6):949-59. doi: 10.1038/ijo.2009.286. Epub 2010 Jan 12. PMID 20065965
- [Background] Weber RV, Buckley MC, Fried SK, Kral JG. Subcutaneous lipectomy causes a metabolic syndrome in hamsters. Am J Physiol Regul Integr Comp Physiol. 2000 Sep;279(3):R936-43. doi: 10.1152/ajpregu.2000.279.3.R936. PMID 10956251
- [Background] Tran TT, Yamamoto Y, Gesta S, Kahn CR. Beneficial effects of subcutaneous fat transplantation on metabolism. Cell Metab. 2008 May;7(5):410-20. doi: 10.1016/j.cmet.2008.04.004. PMID 18460332
- [Background] Elbers JM, Asscheman H, Seidell JC, Gooren LJ. Effects of sex steroid hormones on regional fat depots as assessed by magnetic resonance imaging in transsexuals. Am J Physiol. 1999 Feb;276(2):E317-25. doi: 10.1152/ajpendo.1999.276.2.E317. PMID 9950792
- [Background] Elbers JM, Asscheman H, Seidell JC, Megens JA, Gooren LJ. Long-term testosterone administration increases visceral fat in female to male transsexuals. J Clin Endocrinol Metab. 1997 Jul;82(7):2044-7. doi: 10.1210/jcem.82.7.4078. PMID 9215270
- [Background] Lavebratt C, Almgren M, Ekstrom TJ. Epigenetic regulation in obesity. Int J Obes (Lond). 2012 Jun;36(6):757-65. doi: 10.1038/ijo.2011.178. Epub 2011 Sep 13. PMID 21912396
- [Background] Perrot-Sinal TS. Do these genes make me look fat? Endocrinology. 2009 Mar;150(3):1075-7. doi: 10.1210/en.2008-1586. No abstract available. PMID 19240263
- [Background] Shi H, Seeley RJ, Clegg DJ. Sexual differences in the control of energy homeostasis. Front Neuroendocrinol. 2009 Aug;30(3):396-404. doi: 10.1016/j.yfrne.2009.03.004. Epub 2009 Mar 31. PMID 19341761
- [Background] Barker DJ, Gluckman PD, Godfrey KM, Harding JE, Owens JA, Robinson JS. Fetal nutrition and cardiovascular disease in adult life. Lancet. 1993 Apr 10;341(8850):938-41. doi: 10.1016/0140-6736(93)91224-a. PMID 8096277
- [Background] Barker DJ, Hales CN, Fall CH, Osmond C, Phipps K, Clark PM. Type 2 (non-insulin-dependent) diabetes mellitus, hypertension and hyperlipidaemia (syndrome X): relation to reduced fetal growth. Diabetologia. 1993 Jan;36(1):62-7. doi: 10.1007/BF00399095. PMID 8436255
- [Background] Muhlhausler B, Smith SR. Early-life origins of metabolic dysfunction: role of the adipocyte. Trends Endocrinol Metab. 2009 Mar;20(2):51-7. doi: 10.1016/j.tem.2008.10.006. Epub 2008 Dec 16. PMID 19095460
- [Background] Armitage JA, Khan IY, Taylor PD, Nathanielsz PW, Poston L. Developmental programming of the metabolic syndrome by maternal nutritional imbalance: how strong is the evidence from experimental models in mammals? J Physiol. 2004 Dec 1;561(Pt 2):355-77. doi: 10.1113/jphysiol.2004.072009. Epub 2004 Sep 30. PMID 15459241
- [Background] McMillen IC, Robinson JS. Developmental origins of the metabolic syndrome: prediction, plasticity, and programming. Physiol Rev. 2005 Apr;85(2):571-633. doi: 10.1152/physrev.00053.2003. PMID 15788706
- [Background] Martin RJ, Hausman GJ, Hausman DB. Regulation of adipose cell development in utero. Proc Soc Exp Biol Med. 1998 Dec;219(3):200-10. doi: 10.3181/00379727-219-44333. PMID 9824542
- [Background] Barker M, Robinson S, Osmond C, Barker DJ. Birth weight and body fat distribution in adolescent girls. Arch Dis Child. 1997 Nov;77(5):381-3. doi: 10.1136/adc.77.5.381. PMID 9487954
- [Background] Tchoukalova YD, Nathanielsz PW, Conover CA, Smith SR, Ravussin E. Regional variation in adipogenesis and IGF regulatory proteins in the fetal baboon. Biochem Biophys Res Commun. 2009 Mar 13;380(3):679-83. doi: 10.1016/j.bbrc.2009.01.149. Epub 2009 Jan 29. PMID 19285021
- [Background] Tchoukalova YD, Votruba SB, Tchkonia T, Giorgadze N, Kirkland JL, Jensen MD. Regional differences in cellular mechanisms of adipose tissue gain with overfeeding. Proc Natl Acad Sci U S A. 2010 Oct 19;107(42):18226-31. doi: 10.1073/pnas.1005259107. Epub 2010 Oct 4. PMID 20921416
- [Background] Tchkonia T, Giorgadze N, Pirtskhalava T, Tchoukalova Y, Karagiannides I, Forse RA, DePonte M, Stevenson M, Guo W, Han J, Waloga G, Lash TL, Jensen MD, Kirkland JL. Fat depot origin affects adipogenesis in primary cultured and cloned human preadipocytes. Am J Physiol Regul Integr Comp Physiol. 2002 May;282(5):R1286-96. doi: 10.1152/ajpregu.00653.2001. PMID 11959668
- [Background] Terashima M, Barbour S, Ren J, Yu W, Han Y, Muegge K. Effect of high fat diet on paternal sperm histone distribution and male offspring liver gene expression. Epigenetics. 2015;10(9):861-71. doi: 10.1080/15592294.2015.1075691. PMID 26252449
- [Background] McPherson NO, Owens JA, Fullston T, Lane M. Preconception diet or exercise intervention in obese fathers normalizes sperm microRNA profile and metabolic syndrome in female offspring. Am J Physiol Endocrinol Metab. 2015 May 1;308(9):E805-21. doi: 10.1152/ajpendo.00013.2015. Epub 2015 Feb 17. PMID 25690453
- [Background] Divoux A, Karastergiou K, Xie H, Guo W, Perera RJ, Fried SK, Smith SR. Identification of a novel lncRNA in gluteal adipose tissue and evidence for its positive effect on preadipocyte differentiation. Obesity (Silver Spring). 2014 Aug;22(8):1781-5. doi: 10.1002/oby.20793. Epub 2014 May 23. PMID 24862299
- [Background] Karastergiou K, Fried SK, Xie H, Lee MJ, Divoux A, Rosencrantz MA, Chang RJ, Smith SR. Distinct developmental signatures of human abdominal and gluteal subcutaneous adipose tissue depots. J Clin Endocrinol Metab. 2013 Jan;98(1):362-71. doi: 10.1210/jc.2012-2953. Epub 2012 Nov 12. PMID 23150689
- [Background] Boston RC, Stefanovski D, Moate PJ, Sumner AE, Watanabe RM, Bergman RN. MINMOD Millennium: a computer program to calculate glucose effectiveness and insulin sensitivity from the frequently sampled intravenous glucose tolerance test. Diabetes Technol Ther. 2003;5(6):1003-15. doi: 10.1089/152091503322641060. PMID 14709204
- [Background] Livesey G, Elia M. Estimation of energy expenditure, net carbohydrate utilization, and net fat oxidation and synthesis by indirect calorimetry: evaluation of errors with special reference to the detailed composition of fuels. Am J Clin Nutr. 1988 Apr;47(4):608-28. doi: 10.1093/ajcn/47.4.608. PMID 3281434
- [Background] Shadid S, Koutsari C, Jensen MD. Direct free fatty acid uptake into human adipocytes in vivo: relation to body fat distribution. Diabetes. 2007 May;56(5):1369-75. doi: 10.2337/db06-1680. Epub 2007 Feb 7. PMID 17287467
- [Background] Landt SG, Marinov GK, Kundaje A, Kheradpour P, Pauli F, Batzoglou S, Bernstein BE, Bickel P, Brown JB, Cayting P, Chen Y, DeSalvo G, Epstein C, Fisher-Aylor KI, Euskirchen G, Gerstein M, Gertz J, Hartemink AJ, Hoffman MM, Iyer VR, Jung YL, Karmakar S, Kellis M, Kharchenko PV, Li Q, Liu T, Liu XS, Ma L, Milosavljevic A, Myers RM, Park PJ, Pazin MJ, Perry MD, Raha D, Reddy TE, Rozowsky J, Shoresh N, Sidow A, Slattery M, Stamatoyannopoulos JA, Tolstorukov MY, White KP, Xi S, Farnham PJ, Lieb JD, Wold BJ, Snyder M. ChIP-seq guidelines and practices of the ENCODE and modENCODE consortia. Genome Res. 2012 Sep;22(9):1813-31. doi: 10.1101/gr.136184.111. PMID 22955991
- [Derived] Divoux A, Eroshkin A, Erdos E, Sandor K, Osborne TF, Smith SR. DNA Methylation as a Marker of Body Shape in Premenopausal Women. Front Genet. 2021 Jul 29;12:709342. doi: 10.3389/fgene.2021.709342. eCollection 2021. PMID 34394195
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org